CLINICAL TRIAL: NCT00333619
Title: Non-Pharmacological Interventions on Sleep in Post-Acute Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IIR 04-321
Record Dates: First submitted 2006-06-02; First posted 2006-06-06 (Estimated); Results first posted 2015-04-06 (Estimated); Last update posted 2015-04-24 (Estimated); Status verified 2014-10

CONDITIONS: Sleep Disorders
Keywords: sleep disorders; rehabilitation; rehabilitation outcomes
MeSH Terms: conditions — Sleep Wake Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nonpharmacological sleep intervention (Experimental): The intervention will combine: 1) structured sleep assessment, 2) environmental interventions (efforts to increase bright light exposure, decrease daytime in-bed time, and provide a structured bedtime routine), and 3) elements of cognitive-behavioral strategies.
  Interventions: Behavioral: Nonpharmacological sleep intervention
- Active control (Active Comparator): Daily 15-minute social visit from a research assistant. The visits include structured activities to facilitate social interaction (e.g., memory games, current event discussions).
  Interventions: Behavioral: Active control

INTERVENTIONS:
Behavioral: Nonpharmacological sleep intervention — The intervention combines: 1) structured sleep assessment, 2) environmental interventions (efforts to increase bright light exposure, decrease daytime in-bed time, and provide a structured bedtime routine), and 3) elements of cognitive-behavioral strategies
  Arms: Nonpharmacological sleep intervention
Behavioral: Active control — Daily 15-minute social visit from a research assistant. The visits include structured activities to facilitate social interaction (e.g., memory games, current event discussions).
  Arms: Active control

SUMMARY:
This project is a randomized controlled trial to test whether a multicomponent, nonpharmacological intervention improves sleep/wake patterns and functional recovery among older people undergoing post-acute rehabilitation.

DETAILED DESCRIPTION:
The purpose of this study is to perform a randomized controlled trial to test whether a multicomponent, nonpharmacological intervention improves sleep/wake patterns and functional recovery among older people (N = 214) undergoing post-acute rehabilitation. The intervention will combine: 1) structured sleep assessment, 2) patient education in key elements of cognitive behavioral strategies to improve sleep, and 3) environmental interventions on factors which likely contribute to abnormal sleep/wake patterns in the post-acute rehabilitation setting.

This project will be conducted in a VA post-acute rehabilitation site. Older veterans (>= 60 years) who were previously community-dwelling (N = 214) will be randomized to receive the intervention, or a social contact and memory skills training program as the control condition. Data collected at baseline will include medical data and demographics, as well as subjective and objective measures of sleep, structured assessments of functional status, and medical comorbidity. Follow-up assessments will be performed in the facility while the intervention/control condition is in place, and at three months and six months after discharge from rehabilitation. The main outcome measures will include objective sleep measures (nighttime percent sleep and daytime percent sleep) and functional status collected at three and six months follow-up. Data will be analyzed for all randomized participants in an intention to treat analysis.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged > or = 60, who are admitted to inpatient rehabilitation services, who lived in a non-institutional setting prior to admission, and are admitted for rehabilitation

Exclusion Criteria:

* severe sleep apnea
* severe cognitive impairment
* not enrolled within one week of admission to rehabilitation unit
* too ill to participate
* and planned discharge to a nursing home for total nursing care

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2007-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cathy A. Alessi, MD, Principal Investigator — VA Greater Los Angeles Healthcare System, Sepulveda, CA
Locations (1):
- VA Greater Los Angeles Healthcare System, Sepulveda, CA, Sepulveda, California, United States

REFERENCES:
- [Result] Martin JL, Jouldjian S, Mitchell MN, Josephson KR, Alessi CA. A longitudinal study of poor sleep after inpatient post-acute rehabilitation: the role of depression and pre-illness sleep quality. Am J Geriatr Psychiatry. 2012 Jun;20(6):477-84. doi: 10.1097/JGP.0b013e31824877c1. PMID 22617164
- [Result] Skibitsky M, Edelen MO, Martin JL, Harker J, Alessi C, Saliba D. Can standardized sleep questionnaires be used to identify excessive daytime sleeping in older post-acute rehabilitation patients? J Am Med Dir Assoc. 2012 Feb;13(2):127-35. doi: 10.1016/j.jamda.2010.05.004. Epub 2010 Oct 2. PMID 21450184
- [Result] Martin JL, Dzierzewski JM, Mitchell M, Fung CH, Jouldjian S, Alessi CA. Patterns of sleep quality during and after postacute rehabilitation in older adults: a latent class analysis approach. J Sleep Res. 2013 Dec;22(6):640-7. doi: 10.1111/jsr.12066. Epub 2013 Jul 8. PMID 23834036

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nonpharmacological Sleep Intervention | Active Control
Started | 110 | 109
Post-treatment | 109 | 109
3-month Follow-up | 101 | 105
Completed | 89 | 99
Not Completed | 21 | 10
Not completed — Death | 12 | 6
Not completed — Withdrawal by Subject | 6 | 1
Not completed — Lost to Follow-up | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nonpharmacological Sleep Intervention | Active Control | Total
Number analyzed (Participants) | 110 | 109 | 219
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.39 (9.78) | 73.32 (10.12) | 72.4 (9.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 8
  Male | 105 | 106 | 211
Pittsburgh Sleep Quality Index [Mean (Standard Deviation); unit: units on a scale; 0-21] — The PSQI is a 18-item questionnaire that measures subjective sleep quality and sleep disturbances (total score ranging from 0 - 21; score > 8 indicates poor sleep quality).
  units on a scale; 0-21 | 7.9 (4.1) | 9.2 (4.3) | 8.4 (4.5)
Sleep efficiency [Mean (Standard Deviation); unit: Percentage of time asleep while in bed] — Average sleep efficiency calculated from 7 days of actigraphy. Sleep efficiency for each night is calculated as the number of hours asleep divided by the number of hours in bed.
  Percentage of time asleep while in bed | 70.3 (18.2) | 66.7 (20.2) | 68.6 (19.3)

OUTCOME MEASURES:

1. Primary Outcome: Pittsburgh Sleep Quality Index
Description: The PSQI is a 18-item questionnaire that measures subjective sleep quality and sleep disturbances (total score ranging from 0 - 21; score > 8 indicates poor sleep quality).
Time Frame: 3-month follow-up
Measure: Mean (Standard Deviation); unit: units on a scale; 0-21
Arm/Group | Nonpharmacological Sleep Intervention | Active Control
Number analyzed (Participants) | 110 | 109
units on a scale; 0-21 | 8.6 (3.8) | 9.4 (3.8)
Statistical Analysis 1: Comparison: Nonpharmacological Sleep Intervention vs Active Control; Test type: Superiority or Other; p = 0.10, ANOVA

2. Primary Outcome: Sleep Efficiency
Description: Average sleep efficiency calculated from 7 days of actigraphy. Sleep efficiency for each night is calculated as the number of hours asleep divided by the number of hours in bed.
Time Frame: 3-month follow-up
Measure: Mean (Standard Deviation); unit: percentage of time asleep while in bed
Arm/Group | Nonpharmacological Sleep Intervention | Active Control
Number analyzed (Participants) | 110 | 109
percentage of time asleep while in bed | 77.3 (14.8) | 71.0 (17.6)
Statistical Analysis 1: Comparison: Nonpharmacological Sleep Intervention vs Active Control; Test type: Superiority or Other; p = 0.12, ANOVA

ADVERSE EVENTS:
Time Frame: This was a behavioral sleep education intervention. No medications or devices were tested. Data on adverse events were collected over the entire study period (12-months).
Arm/Group | Nonpharmacological Sleep Intervention | Active Control
Serious Adverse Events (participants affected / at risk) | 0/110 | 0/109
Other Adverse Events (participants affected / at risk) | 0/110 | 0/109

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes